CLINICAL TRIAL: NCT04215653
Title: A Phase 3,Double-blinded, Double Dummy, Positive Drug, Parallel, Randomised Controlled Multicenter Trial to Evaluate Efficacy and Safety of Anaprazole Compared With Rabeprazole in Patients With Duodenal Ulcers.
Brief Title: A Phase 3 Randomised Controlled Trial to Evaluate Efficacy and Safety of Anaprazole in Patients With Duodenal Ulcers.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3571-DU-3001
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-11

CONDITIONS: Duodenal Ulcer，DU
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anaprazole Sodium + Rabeprazole Placebo (Experimental): administered orally once every 30-60 minutes before breakfast for 4 weeks
  Interventions: Drug: Anaprazole Sodium; Drug: Rabeprazole Placebo
- Rabeprazole +Anaprazole Sodium Placebo (Active Comparator): administered orally once every 30-60 minutes before breakfast for 4 weeks
  Interventions: Drug: Rabeprazole; Drug: Anaprazole Sodium Placebo

INTERVENTIONS:
Drug: Anaprazole Sodium — administered orally once every 30-60 minutes before breakfast for 4 weeks
  Arms: Anaprazole Sodium + Rabeprazole Placebo
Drug: Rabeprazole — administered orally once every 30-60 minutes before breakfast for 4 weeks
  Arms: Rabeprazole +Anaprazole Sodium Placebo
Drug: Rabeprazole Placebo — administered orally once every 30-60 minutes before breakfast for 4 weeks
  Arms: Anaprazole Sodium + Rabeprazole Placebo
Drug: Anaprazole Sodium Placebo — administered orally once every 30-60 minutes before breakfast for 4 weeks
  Arms: Rabeprazole +Anaprazole Sodium Placebo

SUMMARY:
A phase 3,double-blinded, double dummy, parallel, non-inferiority, randomised controlled multicenter trial to evaluate efficacy and safety of 4 weeks treatment of Anaprazole 20mg QD compared with rabeprazole 10mg QD in patients with duodenal ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years, male and female
2. Has endoscopic diagnosis of active duodenal ulcer(s) (A1 or A2 stage) within 7 days prior to randomization
3. 1 or 2 ulcers, 3-15 mm in diameter.
4. Signed informed concent form

Exclusion Criteria:

1. Has malignancy ulcer or malignancy ulcer not excluded, compouned ulcer, stress ulcer, esophageal erosion and ulcer, reflux esophagitis, Zollinger-Ellison syndrome.
2. Has esophageal and gastric varices；
3. With severe compliaction, such as pyloric obstruction, bleeding (Forrest I, IIa and IIb) or perforation, and etc；
4. Has gastric ulcer, or has history of inflammatory bowel disease (such as Crohn's disease or ulcerative colitis)；
5. Has undergone surgical resection or partly resection of esophageal, stomach or duodenum；
6. Has used Proton Pump Inhibitors(PPIs) within 5 days prior to randomization, or continuous more than 3 days of use of Proton Pump Inhibitors within 2 weeks prior to randomization；
7. Has been treated with triple or quandruple Helicobacter pylori eradication therapy included PPIs within 28 days prior to randomization；
8. Current use the drugs (such as systemic glucocorticoids, non steroid anti-inflammatory drugs, or anticoagulation drugs) which may induce ulcer or ulceric bleeding or continuous more than 3 days of use the drugs (such as systemic glucocorticoids, non steroid anti-inflammatory drugs, or anticoagulation drugs) within 28 days prior to randomization；
9. Laboratory tests performed in screning stage revealed Alanine aminotransferase (ALT) or aspartate aminotransferase (AST): > 1.5 upper limit of normal (ULN);
10. Laboratory tests performed in screning stage revealed thyroid stimulating hormone (TSH) or free triiodothyronine (FT3) and free thyroxin ( FT4) : > upper limit of normal (ULN)；
11. Woman in pregnancy or lactation period；
12. Plan for pregancy or not willing to contracept with reliable contraception method during study period and within 90 days after the final time of investigational drug administratio；
13. Have alcohol abuse or drug abuse 1 years prior to screening；
14. Has hypersensitivity or allergy to investigatory drug, comparatory drug or related supplements；
15. Has participated or been participating other clinical trials(non-interventional study is excluded)；
16. Has an uncotroled disease, such as has a history of significant central nervous system (CNS), cardiovascular, pulmonary, hepatic, renal, gastrointestinal, or mental or psychological disorders with drug treatment that,in the opinion of the investigator, would not be suitable for participating this clinical trial.
17. Has a history of malignancy or was treated or not treated for malignancy within 5 years before randomization (the participant may be included in the study if he/she has cured cutaneous basal cell carcinoma), no matter if there is evidence for local relapse or metastasis；
18. Laboratory tests performed in screning stage revealed estimated Glomerular filtration rate（eGFR） <80 mL/min/1.73 m2 calculated by Modification of Diet in Renal Disease(MDRD) equation；
19. In the opinion of the investigator, the patients with other situation would not be suitable for participating this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Estimated)
Dates: Start 2020-01-20 (Estimated); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
The endoscopic healing rate of duodenal ulcers at week 4, evaluated by blinded independency central reading. | Treatment of 4 weeks
  The endoscopic ulcer healing rate is defined as the percentage of patients healed (complete healing and significant response) in whom the endoscopic response of duodenal ulcers at week 4 has been evaluated by blinded independency central reading.

SECONDARY OUTCOMES:
The endoscopic healing rate of duodenal ulcers at week 4, evaluated by investigator reading. | Treatment of 4 weeks
  The endoscopic ulcer healing rate is defined as the percentage of patients healed (complete healing and significant response) in whom the endoscopic response of duodenal ulcers at week 4 has been evaluated by investigators.

REFERENCES:
- [Derived] Ni H, Shi J, Hu M, Zhou N, Yang S. Cost-effectiveness analysis of Anaprazole versus Ilaprazole for the treatment of duodenal ulcers in China. Front Pharmacol. 2024 Jun 7;15:1407435. doi: 10.3389/fphar.2024.1407435. eCollection 2024. PMID 38910891
- [Derived] Zhu H, Pan X, Zhang L, Sun H, Fan H, Pan Z, Huang C, Shi Z, Ding J, Wang Q, Du Y, Lyu N, Li Z. Effect and safety of anaprazole in the treatment of duodenal ulcers: a randomized, rabeprazole-controlled, phase III non-inferiority study. Chin Med J (Engl). 2022 Dec 20;135(24):2941-2949. doi: 10.1097/CM9.0000000000002508. PMID 36580650